CLINICAL TRIAL: NCT02457273
Title: An Open-Label, Single-Arm, Two-Stage, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of TLC388 as Second-line Treatment in Subjects With Poorly Differentiated Neuroendocrine Carcinomas
Brief Title: Phase II Study to Evaluate the Efficacy and Safety of TLC388 for Differentiated Neuroendocrine Carcinomas Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1Z14
Record Dates: First submitted 2015-05-04; First posted 2015-05-29 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2018-12

CONDITIONS: Neuroendocrine Carcinomas
Keywords: PDNC(Poorly Differentiated Neuroendocrine Carcinomas); TLC-388 (Lipotecan®)
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — TLC 388

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Assigned Interventions (Experimental): TLC 388
  Interventions: Drug: TLC 388

INTERVENTIONS:
Drug: TLC 388 — 40 mg/m2 of TLC 388, given as a 30 (+3) minute intravenous infusion, on Days 1, 8 and 15 of a 28-day cycle until PD, unacceptable toxicity or consent withdrawal occurs.
  Other Names: Lipotecan®,

SUMMARY:
Title of Study:

An Open-Label, Single-Arm, Two-Stage, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of TLC388 as Second-line Treatment in Subjects with Poorly Differentiated Neuroendocrine Carcinomas

Investigational product:

Lipotecan®*

*Lipotecan® is the trade name of TLC388 HCl, a Topoisomerase I inhibitor)

Phase of development:

Phase II

Number of subjects:

Plan to enroll 44 subjects

Objectives:

Primary objectives:

To determine the objective response rate

Secondary objectives:

To evaluate Disease control rate, Progression free survival, Overall survival, Safety profile and Biomarkers

DETAILED DESCRIPTION:
This is a phase II, open-label, single-arm, two-stage, multicenter study to evaluate the efficacy and safety of Lipotecan® monotherapy in subjects with poorly differentiated neuroendocrine carcinomas. Only those subjects who have failed to first line chemotherapy (Etoposide plus platinum) due to treatment intolerance or radiographic progressive disease (PD), as per RECIST v1.1, are eligible to participate in the study. The scheduled assessments should be performed as identified on a calendar schedule, and should not be affected by delays in therapy, drug holidays or any other events that might be lead to imbalance in a treatment arm in the timing of disease assessment. Efficacy results are based on radiographic assessments reviewed by the investigator.

Eligible subjects will receive 40 mg/m2 of Lipotecan®, given as a 30 (+3) minute intravenous infusion, on Days 1, 8 and 15 of a 28-day cycle until PD, unacceptable toxicity or consent withdrawal occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed poorly differentiated neuroendocrine carcinomas.
2. Patients who had first-line treatment failure (First line therapy must be etoposide plus platinum) due to treatment intolerance or radiographic progressive disease (as per RECIST v1.1).
3. At least one measurable lesion in a non-irradiated area.
4. Aged > 20 years old.
5. ECOG Performance Status ≤ 2.
6. Life expectancy greater than 12 weeks.
7. Adequate bone marrow function :

   * absolutely neutrophil count ≥ 1500 /mm3 or WBC ≥ 4000/mm3
   * Hemoglobin > 9 g/dl
   * platelet count ≥ 100,000 /mm3
8. Adequate liver function :

   * ALT & AST ≤ 2.5 x ULN if without liver metastasis or ≤ 5 x ULN if with hepatic metastasis Alkaline phosphatase ≤ 2.5 x ULN if without liver and bone metastasis; or ≤ 5 x ULN if with hepatic metastasis or bone metastasis
   * Total Bilirubin < 2 x ULN
9. Adequate renal function: creatinine < 1.5 x ULN.
10. Subjects who are willing and able to comply with all of the study procedures, and able to sign the informed consent.

Exclusion Criteria:

1. Major surgery within two weeks prior to entering the study.
2. Patients with CNS metastasis, including clinical suspicion.
3. Patients who are under active or uncontrolled infections.
4. Patients with concomitant illness that might be aggravated by chemotherapy.
5. Patients who are pregnant or with breast feeding.
6. Other concomitant or previously malignancy within 5 yrs except for in situ cervix cancer or squamous cell carcinoma of the skin treated by surgery only.
7. Fertile men and women unless using a reliable and appropriate contraceptive method
8. A history of or the presence of one or more cardiac diseases, such as congestive heart failure (New York Heart Association Class III or IV), myocardial infarction or unstable angina and related surgeries, within 3 months prior to the initiation of the treatment dose.
9. Patients with a known history of human immunodeficiency virus infection.
10. The presence of active or uncontrolled systemic infection (bacterial, viral, other) except for chronic hepatitis B and hepatitis C.
11. Use of any investigational agent within 4 weeks of baseline.
12. Uncontrolled and unstable concurrent medical or psychiatric illness that will jeopardize the safety of the subject, interfere with the objectives of the protocol, or affect the subject compliance with study requirements, as determined by the investigator.
13. Known hypersensitivity or adverse drug reactions to Lipotecan® or its components.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-07-04 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
the objective response rate | 5 years
  Analysis for the objective response rate will be conducted on both the per protocol(PP) and evaluable data sets.

SECONDARY OUTCOMES:
Disease control rate | 5 years
  The Disease control rate (DCR) is the percentage of subjects who have a best-response rating of CR or PR or SD (DCR= CR+PR+SD) (according to RECIST v1.1) when assessed after every 8 weeks of study drug (up to 6 cycles) and maintained for at least 28 days.
Progression free survival | 5 years
  Progression-free survival will be calculated as the duration between the first date of randomization and the date of disease recurrence or progression according to RECIST v1.1 (failed), taking the status of tumor at the treatment has been completed as the reference, or death (failed), or the date of withdrawal (last contact date, censored), or the scheduled data analysis date (censored).
Overall survival | 5 years
  Overall survival will be calculated from the date of randomization to either the date of death from all causes, or to the date of withdrawal (last contact date, censored), or to the scheduled data analysis date (censored).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 5 years
  Physical examinations, lab abnormality and other toxicities graded by the NCI Common Toxicity Criteria will be examined to evaluate safety profiles of the study treatments. Particular attention will be paid to Grade 3 or 4 toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Chao, MD., PhD, Study Chair — Taipei Veterans General Hospital, Taiwan; Hui-Jen Tsai, MD., PhD, Study Director — National Health Research of Institutes; Ming-Huang Chen, MD., PhD, Study Director — Taipei Veterans General Hospital, Taiwan; Jen-Shi Chen, MD, Principal Investigator — Chang Gung Memorial Hospital; Cheng-Chung Wu, MS, Principal Investigator — Taichung Veterans General Hospital; Chiun Hsu, MD., PhD, Principal Investigator — National Taiwan University Hospital; Chia-Jui Yen, MD., PhD, Principal Investigator — National Cheng-Kung University Hospital; Yen-Yang Chen, MD, Principal Investigator — Chang Gung Memorial Hospital; Ta-Chih Liu, MD., PhD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (7):
- Taiwan (7):
  - Chung Gung Memorial Hospital(Kaohsiung City), Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital (Lin-Kou),, Linkou District
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen MH, Chou WC, Hsiao CF, Jiang SS, Tsai HJ, Liu YC, Hsu C, Shan YS, Hung YP, Hsich CH, Chiu CH, Liu TC, Cho SF, Liu TW, Chao Y. An Open-Label, Single-Arm, Two-Stage, Multicenter, Phase II Study to Evaluate the Efficacy of TLC388 and Genomic Analysis for Poorly Differentiated Neuroendocrine Carcinomas. Oncologist. 2020 May;25(5):e782-e788. doi: 10.1634/theoncologist.2019-0490. Epub 2019 Dec 18. PMID 31852810